CLINICAL TRIAL: NCT06173102
Title: Treatment Effectiveness of Cranial Orthosis Therapy in the Correction of Deformational Plagiocephaly: a Randomized Controlled Pilot Study Comparing Cranial Orthosis Therapy to the Natural Course
Brief Title: Cranial Orthosis Therapy for Plagiocephaly: an RCT Pilot Study Comparing Cranial Orthosis to the Natural Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Camille Costa, Associate Researcher, St. Justine's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2024-5800
Record Dates: First submitted 2023-11-30; First posted 2023-12-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Plagiocephaly; Plagiocephaly, Nonsynostotic; Plagiocephaly, Positional
MeSH Terms: conditions — Plagiocephaly; Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Intervention Model Description: randomization sequence will be created using Microsoft Excel 2022 with a 1:1 allocation using random block sizes of 2 and
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Cranial Orthosis (Experimental): Early cranial orthosis (reception 1 week after initial visit)
  Interventions: Device: Cranial Orthosis
- Usual Cranial Orthosis (Other): Usual cranial orthosis (reception 7 weeks after initial visit)
  Interventions: Device: Cranial Orthosis

INTERVENTIONS:
Device: Cranial Orthosis — Early versus usual reception of orthosis.

SUMMARY:
Our study aims to assess the feasibility of a randomized controlled trial that investigates the efficacy of cranial orthosis therapy for treating severe deformational plagiocephaly in infants between 4 and 7 months old.

The main question it aims to answer are:

• Feasibility of conducting the study in our physiatry clinic.

Participants will be randomized into two groups, receiving cranial orthosis at 1 week post initial visit, or the standard of care (7 weeks post initial visit). They will have head measurements and helmet adjustments as well as medical follow-up with a total of 4 visits. Post-treatment questionnaires will be filled out.

DETAILED DESCRIPTION:
Our research endeavors to examine the feasibility of implementing a randomized controlled trial (RCT) that evaluates the efficacy of cranial orthosis therapy in addressing severe deformational plagiocephaly among infants aged 4 to 7 months.

Primary Objective: The central focus is on evaluating the feasibility aspects associated with the RCT design within our clinical setting.

Participants: Infants meeting the inclusion criteria will be recruited and randomized into two distinct groups:

1. Treatment Group: Receiving cranial orthosis therapy initiated one week post their initial physiatrist visit.
2. Control Group: Adhering to the standard of care, with cranial orthosis initiation at 7 weeks post their initial physiatrist visit.

Study Procedures: Participants in both groups will undergo a structured series of assessments and interventions, including:

* Head measurements and 3D-scan evaluations to quantify cranial deformities.
* Helmet adjustments by experienced orthotists based on growth and changes in head shape.
* Regular medical follow-ups, totaling four visits during the course of the study.

Post-Treatment Assessments: Upon completion of the cranial orthosis therapy, participants will be required to fill out post-treatment questionnaires, providing valuable insights into their experiences, satisfaction levels, and any potential concerns

ELIGIBILITY:
Inclusion Criteria:

* All participants must be assessed by a physiatrist at Sainte-Justine Hospital at the plagiocephaly clinic of the physical medicine and rehabilitation service.
* Participants must have a clinical diagnosis of severe deformational plagiocephaly by a physiatrist based on clinical evaluation and confirmed by anthropometric measurements with a spreading caliper and 3D-scan.
* Participants must be aged from 4 months and 0 days to 7 months old minus a day at the onset of cranial orthosis therapy. Premature subjects will be age-adjusted by calculating the post-partum age minus the number of weeks of prematurity, rounding to the whole nearest month.
* Participants' parents (or legal guardian) must be apt to give consent and able to reliably express themselves (either written or verbally, if illiterate or unable to write for any other reason).

Exclusion Criteria:

* Patients whose 3D-scan measurements do not confirm a severe plagiocephaly.
* Participants who are lost at follow-up or who drop out of treatment will be excluded.
* Participants whose parents report less than 20 hours per day on average of helmet wear.
* Participants with synostotic cranial deformation.
* Patients with isolated brachycephaly, without a plagiocephalic component to the deformation.
* Patients with other craniofacial deformities or syndromes.
* Patients having had their orthosis made or modified at a laboratory other than the Sainte-Justine hospital/Centre de réadaptation Marie-Enfant.

Ages: 122 Days to 212 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Qualitative information on Feasibility | through study completion, average of 12 weeks per patient
  documenting difficulties encountered during the pilot study, including but not limited to loss at follow-up, missed appointments, missing questionnaires, difficulties with enrollment, and coordination of appointments between the PM&R service and the Orthotics clinic.

SECONDARY OUTCOMES:
Cranial Vault Asymmetry (CVA) | at week 0, week 6 and week 12
  The difference between the longest and shortest cranial diagonals, measured in millimeters.
Cranial Vault Asymmetry Index (CVAI) | at week 0, week 6 and week 12
  A percentage value that considers the overall size of the head in relation to CVA.
Parental Satisfaction: | through completion of study, on average 12 weeks per patient
  Measured with a parental questionnaire at the end of treatment, assessing satisfaction with head shape and cranial orthosis therapy.
Adverse Effects: | through completion of study, on average 12 weeks per patient
  Any adverse effects observed during cranial orthosis therapy will be collected from parental questionnaires and medical chart records.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Costa, MD, Principal Investigator — Université de Montréal, CHU Sainte-Justine
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No